CLINICAL TRIAL: NCT04990297
Title: Cardiac Magnetic Resonance for Risk Stratification in Dilated Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, Vice Director of Magnetic Resonance Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CREATE
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Dilated Cardiomyopathy; Single-center Study
Keywords: dilated cardiomyopathy; cardiovascular magnetic resonance imaging; prognosis
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — data of radiology imaging, clinical study and laboratory study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dilated cardiomyopathy (DCM) is an increasingly recognized cause of morbidity and mortality with heterogenous etiologies (eg, genetic, environment) and clinical manifestations, characterized by left ventricular (LV) systolic dysfunction and LV or biventricular dilation. Previous publications reported the three-year treated mortality rates remain high at 12%-20% and a reported 5-year mortality rate up to 50%, with death resulting from ventricular arrhythmia leading to sudden cardiac death (SCD) or advanced heart failure (HF). With large fields of view and high spatial resolution, Cardiac magnetic resonance (CMR) is the reference standard for assessing cardiac mass, volume, and function. CMR also provides non noninvasive characterization of the myocardium benefiting to differential diagnosis and risk stratification.

ELIGIBILITY:
Inclusion Criteria:

1. reduced left ventricular ejection fraction (LVEF<50%)
2. LV end-diastolic volume >2SD from normal according to normograms corrected by body surface area (BSA) and age.

Exclusion Criteria:

1. Any evidence indicating the presence of ischemic heart disease:

   Coronary angiography, perfusion imaging Medical documentation that indicated the presence of ischemic heart disease An infarct pattern of late gadolinium enhancement on cardiac magnetic resonance studies and/or acute coronary syndrome or coronary revascularization during follow-up
2. Any evidence of hypertrophic cardiomyopathy, or moderate-to-severe valvular disease[18], or infiltrative disease (such as amyloidosis, sarcoidosis, Fabry disease)
3. Incessant arrhythmias
4. Inability to lie flat
5. Pregnancy
6. Contraindication to cardiac magnetic resonance including severe claustrophobia, defibrillators, pacemakers, certain types of intracranial aneurysm clips, intraocular metal, and Stage IV/V chronic kidney disease
7. Diabetes mellitus with end organ damage
8. Inability to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a prospective, single-center, observational registry including consecutive patients with DCM who undergo clinical evaluation, blood draw for genetics and biomarker assessment, echocardiography, and CMR.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-12-24 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause Mortality | 1-10years
  the incidence of all-cause death the incidence of all-cause death the incidence of all-cause death the incidence of all-cause mortality

SECONDARY OUTCOMES:
A composite of SCD and aborted SCD | 1-10years
  SCD, defined as unexpected death within ≤1 hour of cardiac symptoms in the absence of any progressive cardiac deterioration, during sleep, or ≤24 hours of last being seen alive. Aborted SCD, defined as an appropriate implantable cardioverter defibrillator shock for ventricular arrhythmia, a nonfatal episode of ventricular fibrillation or spontaneous sustained ventricular tachycardia causing hemodynamic compromise and requiring cardioversion
Deterioration of HF | 1-10years
  HF-death, heart transplantation, left ventricular assist device
Major adverse cardiac events | 1-10years
  all-cause mortality, heart transplantation, left ventricular assist device, aborted SCD, sustained ventricular tachycardia and hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Minjie Lu, PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Our study data is applicable to other researchers with permmsion.

REFERENCES:
- [Result] Shah KS, Xu H, Matsouaka RA, Bhatt DL, Heidenreich PA, Hernandez AF, Devore AD, Yancy CW, Fonarow GC. Heart Failure With Preserved, Borderline, and Reduced Ejection Fraction: 5-Year Outcomes. J Am Coll Cardiol. 2017 Nov 14;70(20):2476-2486. doi: 10.1016/j.jacc.2017.08.074. Epub 2017 Nov 12. PMID 29141781
- [Result] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Result] Stecker EC, Vickers C, Waltz J, Socoteanu C, John BT, Mariani R, McAnulty JH, Gunson K, Jui J, Chugh SS. Population-based analysis of sudden cardiac death with and without left ventricular systolic dysfunction: two-year findings from the Oregon Sudden Unexpected Death Study. J Am Coll Cardiol. 2006 Mar 21;47(6):1161-6. doi: 10.1016/j.jacc.2005.11.045. Epub 2006 Feb 23. PMID 16545646
- [Result] Rahimi K, Bennett D, Conrad N, Williams TM, Basu J, Dwight J, Woodward M, Patel A, McMurray J, MacMahon S. Risk prediction in patients with heart failure: a systematic review and analysis. JACC Heart Fail. 2014 Oct;2(5):440-6. doi: 10.1016/j.jchf.2014.04.008. Epub 2014 Sep 3. PMID 25194291
- [Result] Fukushima A, Milner K, Gupta A, Lopaschuk GD. Myocardial Energy Substrate Metabolism in Heart Failure : from Pathways to Therapeutic Targets. Curr Pharm Des. 2015;21(25):3654-64. doi: 10.2174/1381612821666150710150445. PMID 26166604
- [Result] Marwick TH, Shah SJ, Thomas JD. Myocardial Strain in the Assessment of Patients With Heart Failure: A Review. JAMA Cardiol. 2019 Mar 1;4(3):287-294. doi: 10.1001/jamacardio.2019.0052. PMID 30810702
- [Result] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455
- [Result] Gormeli CA, Ozdemir ZM, Kahraman AS, Yagmur J, Ozdemir R, Colak C. The evaluation of non-ischemic dilated cardiomyopathy with T1 mapping and ECV methods using 3T cardiac MRI. Radiol Med. 2017 Feb;122(2):106-112. doi: 10.1007/s11547-016-0701-y. Epub 2016 Oct 27. PMID 27785679
- [Result] Barison A, Del Torto A, Chiappino S, Aquaro GD, Todiere G, Vergaro G, Passino C, Lombardi M, Emdin M, Masci PG. Prognostic significance of myocardial extracellular volume fraction in nonischaemic dilated cardiomyopathy. J Cardiovasc Med (Hagerstown). 2015 Oct;16(10):681-7. doi: 10.2459/JCM.0000000000000275. PMID 26090916
- [Result] Inui K, Asai K, Tachi M, Yoshinaga A, Izumi Y, Kubota Y, Murai K, Tsukada YT, Amano Y, Kumita S, Shimizu W. Extracellular volume fraction assessed using cardiovascular magnetic resonance can predict improvement in left ventricular ejection fraction in patients with dilated cardiomyopathy. Heart Vessels. 2018 Oct;33(10):1195-1203. doi: 10.1007/s00380-018-1154-0. Epub 2018 Mar 20. PMID 29560528
- [Result] Vita T, Grani C, Abbasi SA, Neilan TG, Rowin E, Kaneko K, Coelho-Filho O, Watanabe E, Mongeon FP, Farhad H, Rassi CH, Choi YL, Cheng K, Givertz MM, Blankstein R, Steigner M, Aghayev A, Jerosch-Herold M, Kwong RY. Comparing CMR Mapping Methods and Myocardial Patterns Toward Heart Failure Outcomes in Nonischemic Dilated Cardiomyopathy. JACC Cardiovasc Imaging. 2019 Aug;12(8 Pt 2):1659-1669. doi: 10.1016/j.jcmg.2018.08.021. Epub 2018 Nov 15. PMID 30448130